CLINICAL TRIAL: NCT01646320
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Therapy With Dapagliflozin Added to Saxagliptin in Combination With Metformin Compared to Therapy With Placebo Added to Saxagliptin in Combination With Metformin in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Metformin and Saxagliptin
Brief Title: Safety and Efficacy of Dapagliflozin in Triple Therapy to Treat Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB102-129; 2011-006324-20 (EudraCT Number)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; saxagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1: Dapagliflozin (10 mg) + Saxagliptin + Metformin IR (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Saxagliptin; Drug: Metformin immediate release (IR)
- Arm 2: Placebo + Saxagliptin + Metformin IR (Experimental)
  Interventions: Drug: Placebo matching with Dapagliflozin; Drug: Saxagliptin; Drug: Metformin immediate release (IR)

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 10 mg, Once daily, Up to 52 weeks
  Arms: Arm1: Dapagliflozin (10 mg) + Saxagliptin + Metformin IR
Drug: Placebo matching with Dapagliflozin — Tablets, Oral, 0 mg, Once daily, Up to 52 weeks
  Arms: Arm 2: Placebo + Saxagliptin + Metformin IR
Drug: Saxagliptin — Tablets, Oral, 5 mg, Once daily, Up to 52 weeks
  Other Names: Onglyza
Drug: Metformin immediate release (IR) — Tablets, Oral, ≥ 1500 mg, Twice daily, Up to 52 weeks

SUMMARY:
The purpose of this study is to learn if BMS-512148 (Dapagliflozin) as part of a triple combination therapy can improve (decrease) hemoglobin A1c in patients with type 2 diabetes after 24 weeks of treatment compared to a 2 drug oral antidiabetic therapy. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Prior to randomization, all eligible subjects will receive open-label treatment with Saxagliptin 5mg and Metformin IR during the 16-week open-label treatment period.

ELIGIBILITY:
Inclusion Criteria

1. Signed Written Informed Consent

   1. Subjects must be willing and able to give signed and dated written informed consent.
2. Target Population

   For inclusion into Stratum A:

   i) Subjects with T2DM with inadequate glycemic control, defined as central laboratory HbA1c ≥ 8.0 and ≤ 11.5% obtained at the screening visit (ie Week -18 visit), on stable metformin therapy alone for at least 8 weeks prior to screening visit at a dose ≥ 1500 mg per day

   For inclusion into Stratum B:

   ii) Subjects with T2DM with inadequate glycemic control, and HbA1c ≥ 7.5 and ≤ 10.5% obtained at the screening visit and on stable metformin therapy at a dose ≥ 1500 mg per day AND a DPP4 inhibitor at the maximum approved dose for at least 8 weeks prior to screening visit.

   b) C-peptide ≥ 1.0 ng/mL (0.34 nmol/L) at screening visit. c) BMI ≤ 45.0 kg/m2 at the screening visit.
3. Age and Reproductive Status

   1. Men and women, aged ≥ 18 years old at time of screening visit.
   2. Women of childbearing potential (WOCBP) must be using an acceptable method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized.
   3. WOCBP must have a negative serum or urine pregnancy test within 24 hours prior to the start of investigational product.
   4. Women must not be breastfeeding
   5. Sexually active fertile men must use highly effective birth control if their partners are WOCBP.

Exclusion Criteria

1. Target Disease Exceptions

   1. History of diabetes insipidus
   2. Symptoms of poorly controlled diabetes that would preclude participation in this trial including but not limited to marked polyuria and polydipsia with greater than 10% weight loss during the three months prior to screening, or other signs and symptoms.
   3. History of diabetic ketoacidosis or hyperosmolar nonketotic coma.
2. Medical History and Concurrent Diseases

   1. History of bariatric surgery or lap-band procedure within 12 months prior to screening.
   2. Any unstable endocrine, psychiatric or rheumatic disorders as judged by the Investigator.
   3. Subject who, in the judgment of the investigator, may be at risk for dehydration or volume depletion that may affect the interpretation of efficacy or safety data and concomitant use of loop diuretics in countries where this is not recognized in the Dapagliflozin label.
   4. Subject is currently abusing alcohol or other drugs or has done so within the last 6 months.

      Acute Vascular Event:
   5. Uncontrolled hypertension defined as systolic blood pressure (SBP) ≥ 160 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg.
   6. Cardiovascular Disease within 3 months of the screening visit [ie myocardial infarction, cardiac surgery or revascularization (CABG/PTCA), unstable angina, stroke or transient ischemic attack (TIA)].
   7. Congestive heart failure as New York Association (NYHA) class IV, unstable or acute congestive heart failure.

      Renal Diseases:
   8. Moderate or severe impairment of renal function [defined as eGFR < 60 mL/min/1.73m2 (estimated by MDRD) or serum creatinine (Scr) ≥ 1.5 mg/dL in males or ≥ 1.4 mg/dL in females.]
   9. Conditions of congenital renal glucosuria

      Hepatic Diseases:
   10. Significant hepatic disease, including, but not limited to, chronic active hepatitis and/or severe hepatic insufficiency, including subjects with ALT and/or AST > 3x ULN and or Total Bilirubin > 2.5 x ULN.

       Hematological and Oncological Disease/Conditions:
   11. History of hemoglobinopathy, with the exception of sickle cell trait (SA) or thalassemia minor; or chronic or recurrent hemolysis.
   12. Malignancy within 5 years of the screening visit (with the exception of treated basal cell or treated squamous cell carcinoma)
   13. Known immunocompromised status, including but not limited to, individuals who have undergone organ transplantation or who are positive for the human immunodeficiency virus.
   14. Donation of blood or blood products to a blood bank, blood transfusion, or participation in a clinical study requiring withdrawal of > 400 mL of blood during the 6 months prior to the screening visit.

       Prohibited treatment and therapies:
   15. Administration of any antihyperglycemic therapy, other than metformin and DPP4's, for more than 14 days (consecutive or not) during the 12 weeks prior to screening, as well as previous exposure to DPP4 or SGLT-2 inhibitor in any DPP4 or SGLT-2 inhibitor trial is an exclusion criterion.
   16. Current treatment with potent cytochrome P450 3A4/5 inhibitors (in countries where dose adjustment would be required by the dapagliflozin label).
   17. Administration of any other investigational drug or participation in any interventional clinical studies within 30 days of planned screening to this study. Subjects who failed to satisfy all eligibility criteria at screening and did not enter the lead-in or open-label period in CV181-168 or CV181-169 studies specifically, do not need to wait 30 days.
3. Physical and Laboratory Test Findings

   a) Hemoglobin ≤ 11.0 g/dL (110 g/L) for men; hemoglobin ≤ 10.0 g/dL (100 g/L) for women

   b) Presence of hematuria:

   i) For male subjects being considered for Stratum A: microscopic hematuria present at Week -18 or Week -16 AND no common cause that can be confirmed is exclusionary. Male subjects with a confirmed common cause can be entered into the open-label phase with a documented negative result for hematuria microscopic urinalysis performed by the central laboratory.

   ii) For male subjects being considered for Stratum B: microscopic hematuria present at Week -10 or Week -8 AND no common cause that can be confirmed is exclusionary. Male subjects with a confirmed common cause can be entered into the open-label phase with a documented negative result for hematuria microscopic urinalysis performed by the central laboratory.

   NOTE: Female sub}ects with hematuria can be entered into the open-label phase and be randomized, but should be investigated according to local standards and best clinical practices. (See Appendix 3)

   c) Other central laboratory test findings:

   - Abnormal free T4 values. Abnormal thyroid stimulating hormone (TSH) value at screening will be further evaluated by free T4. Sub}ects with abnormal free T4 values will be excluded.
   * Positive for hepatitis B surface antigen
   * Positive for anti-hepatitis C virus antibody
4. Allergies and Adverse Drug Reaction

   a) Subjects who have contraindications to therapy as outlined in the dapagliflozin and saxagliptin Investigator Brochure, the local dapagliflozin or saxagliptin package insert or the local metformin package insert, including current treatment with potent cytochrome P450 3A4/5 inhibitors (in countries where dose adjustment would be required by the local Onglyza (saxagliptin) label.
5. Sex and Reproductive Status

   a) Women who are pregnant
6. Other Exclusion Criteria

   1. Prisoners or subjects who are involuntarily incarcerated
   2. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
   3. Subjects on a commercial weight loss program with ongoing weight loss, or on an intensive exercise program.
   4. Employee of BMS, AstraZeneca (AZ), or their relatives.
   5. Subject with any condition which, in the judgment of the Investigator, may render the subject unable to complete the study or which may pose a significant risk to the subject.
   6. Subject is a participating investigator, study coordinator, employee of an investigator or immediate family member of any of the aforementioned.

      Open Label Treatment Period

      Note: Enrollment of subjects into the open-label (Stratum A) treatment period, beginning eee -16 of the study with HbA1c values at the lower bound (≥ 8.0% and ≤ 9.0%) and Enrollment of subjects into the open-label (Stratum B) eee -8, of the study with HbA1c values at the lower bound (≥ 7.5% and ≤ 8.5%) will be limited to approximately 50% of the total number of subjects randomized.

      • For subject in Stratum A:
      * At Week -10 and Week -2 a FPG qualification check will be performed. Subjects with a central laboratory FPG value meeting > 270 mg/dL will be scheduled for a follow-up visit (within 3 - 5 days) to obtain a second central laboratory FPG value. If the mean of the originally scheduled central laboratory FPG and the repeat central laboratory FPG value is > 270 mg/dL, the subject cannot be randomized and must be discontinued.

        * For subjects in Stratum B:
      * At Week -2 a FPG qualification check will be performed. Subjects with a central laboratory FPG value meeting > 270 mg/dL will be scheduled for a follow-up visit (within 3 - 5 days) to obtain a second central laboratory FPG value. If the mean of the originally scheduled central laboratory FPG and the repeat central laboratory FPG value is > 270 mg/dL, the subject cannot be randomized and must be discontinued

      Double Blind Treatment Period

      Inclusion criteria:

      • For Stratum A AND Stratum B:

      - Subjects with T2DM with inadequate glycemic control, defined as central laboratory HbA1c ≥ 7.0 and ≤ 10.5% obtained at the Week -2 visit of the open-label treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (56):
- United States (26):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Clinical Research Advantage Inc/Desert Clinical Research Llc, Mesa, Arizona
  - Clinical Research Advantage, Inc., Phoenix, Arizona
  - Elite Clinical Studies, Llc, Phoenix, Arizona
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Randall G. Shue, Do, Inc., Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Diabetes Medical Center Of California, Northridge, California
  - Cassidy Medical Group/Clinical Research Advantage, Vista, California
  - Palm Springs Research Institute, Hialeah, Florida
  - Fpa Clinical Research, Kissimmee, Florida
  - International Research Associates, Llc, Miami, Florida
  - Omega Research Consultants, Llc, Orlando, Florida
  - Compass Research East, Llc, Oviedo, Florida
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - Cedar Crosse Research Center, Chicago, Illinois
  - Clinical Research Advantage, Evansville, Indiana
  - Associated Internal Medicine Specialists, Battle Creek, Michigan
  - Jackson Clinic, Rolling Fork, Mississippi
  - Premier Research, Trenton, New Jersey
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - Sterling Research Grp, Ltd., Cincinnati, Ohio
  - Endocrine Associates, Houston, Texas
  - Sam Clinical Research Center, San Antonio, Texas
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
- Czechia (4):
  - Local Institution, Broumov
  - Local Institution, Pardubice
  - Local Institution, Prague
  - Local Institution, Pribram V
- Mexico (4):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Monterrey, Nuevo León
- Poland (5):
  - Local Institution, Bialystok
  - Local Institution, Krakow
  - Local Institution, Ruda Śląska
  - Local Institution, Warsaw
  - Local Institution, Żory
- Clinical Research Puerto Rico, San Juan, Puerto Rico
- Romania (6):
  - Local Institution, Bucharest, Bucharest
  - Local Institution, Bucharest
  - Local Institution, Constanța
  - Local Institution, Craiova
  - Local Institution, Galati
  - Local Institution, Ploieşti
- Russia (4):
  - Local Institution, Kursk
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Yaroslaval
- United Kingdom (6):
  - Local Institution, Portsmouth, Hants
  - Local Institution, Newport, Isle of Wight
  - Local Institution, Liverpool, Merseyside
  - Local Institution, Chippenham, Wiltshire
  - Local Institution, Bedfordshire
  - Local Institution, London

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Mathieu C, Catrinoiu D, Ranetti AE, Johnsson E, Hansen L, Chen H, Garcia-Sanchez R, Iqbal N, Celinski A. Characterization of the Open-Label Lead-In Period of Two Randomized Controlled Phase 3 Trials Evaluating Dapagliflozin, Saxagliptin, and Metformin in Type 2 Diabetes. Diabetes Ther. 2018 Aug;9(4):1703-1711. doi: 10.1007/s13300-018-0445-x. Epub 2018 May 25. PMID 29802530
- [Derived] Mathieu C, Ranetti AE, Li D, Ekholm E, Cook W, Hirshberg B, Chen H, Hansen L, Iqbal N. Randomized, Double-Blind, Phase 3 Trial of Triple Therapy With Dapagliflozin Add-on to Saxagliptin Plus Metformin in Type 2 Diabetes. Diabetes Care. 2015 Nov;38(11):2009-17. doi: 10.2337/dc15-0779. Epub 2015 Aug 5. PMID 26246458
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Trial with Dapagliflozin added to Saxagliptin in Combination with Metformin compared to placebo added to Saxagliptin in combination with Metformin in Subjects with Type 2 Diabetes who have Inadequate Glycemic Control on Metformin and Saxagliptin
Pre-assignment Details: Arm1: Dapagliflozin (10 mg) + Saxagliptin + Metformin IR
  Arm 2: Placebo + Saxagliptin + Metformin IR
Groups:
- Dapa+Saxa+Met: Participants received dapagliflozin, 10 mg, and open-label saxagliptin 5 mg and metformin ≥1500 mg per day for up to 52 weeks
- Pla+Saxa+Met: Participants received dapagliflozin matching placebo and open-label saxagliptin 5 mg and metformin ≥1500 mg per day for up to 52 weeks
Period: Short-term Period (Day 1 to Week 24)
Arm/Group | Dapa+Saxa+Met | Pla+Saxa+Met
Started | 160 | 160
Completed | 148 | 153
Not Completed | 12 | 7
Not completed — Adverse Event | 3 | 0
Not completed — No longer meets study criteria | 0 | 1
Not completed — Not reported | 2 | 2
Not completed — Other | 1 | 0
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 2 | 0
Period: Long-term Period (Weeks 24 to 52)
Arm/Group | Dapa+Saxa+Met | Pla+Saxa+Met
Started | 147 | 147
Completed | 141 | 140
Not Completed | 6 | 7
Not completed — Subject no longer meets study criteria | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 4 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized subjects who received at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapa+Saxa+Met | Pla+Saxa+Met | Total
Number analyzed (Participants) | 160 | 160 | 320
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 55.2 (8.61) | 55.0 (9.60) | 55.1 (9.10) [30 to 75]
Age, Customized [Number; unit: Participants]
  < 65 years | 137 | 132 | 269
  >= 65 years | 23 | 28 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 84 | 174
  Male | 70 | 76 | 146
Race/Ethnicity, Customized [Number; unit: Participants]
  ASIAN | 1 | 1 | 2
  BLACK/AFRICAN AMERICAN | 8 | 10 | 18
  OTHER | 1 | 2 | 3
  WHITE | 150 | 147 | 297
  AMERICAN INDIAN/ALASKA NATIVE | 0 | 0 | 0
  NATIVE HAWAIIAN/OTHER PACIFIC ISLANDER | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) at Week 24
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 6, 12, 18, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: The Randomized Subjects Data Set consists of all randomized subjects who received at least one dose of double-blind study medication during the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: Percentage of glycosylated hemoglobin
Arm/Group | Dapa+Saxa+Met | Pla+Saxa+Met
Number analyzed (Participants) | 158 | 158
Percentage of glycosylated hemoglobin | -0.82 (0.0686) | -0.1 (0.0704)
Statistical Analysis 1: Comparison: Dapa+Saxa+Met vs Pla+Saxa+Met; Test type: Superiority or Other; p < 0.0001, Longitudinal Repeated Measures Analysis — Tested at alpha=0.05; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-0.91 to -0.53], Standard Error of Mean 0.0964

2. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose at Week 24
Description: Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. FPG measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 6, 12, 18, and 24 in the double-blind period
Time Frame: From Baseline to Week 24
Population: The Randomized Subjects Data Set consists of all randomized subjects who received at least one dose of double-blind study medication during the double-blind treatment period. Number of participants analyzed corresponds to the number of randomized subjects with non-missing baseline value and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapa+Saxa+Met | Pla+Saxa+Met
Number analyzed (Participants) | 158 | 157
mg/dL | -32.7 (2.821) | -5.3 (2.968)
Statistical Analysis 1: Comparison: Dapa+Saxa+Met vs Pla+Saxa+Met; Test type: Superiority or Other; p < 0.0001, Longitudinal Repeated Measures Analysis — Secondary end points are tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -27.5, 95% CI 2-sided [-35.4 to -19.6], Standard Error of Mean 4.015

3. Secondary Outcome: Adjusted Mean Change From Baseline in 120-minute Postprandial Glucose (PPG) at Week 24
Description: 2-hour postprandial glucose (PPG) from a liquid meal tolerance test (2-h MTT) Subject must be fasted for at least 8 hrs prior to the MTT.
Time Frame: From Baseline to Week 24
Population: The Randomized Subjects Data Set consists of all randomized subjects who received at least one dose of double-blind study medication during the double-blind treatment period. Number of participants analyzed is the number of randomized subjects with non-missing baseline and Week 24 (LOCF) values.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dapa+Saxa+Met | Pla+Saxa+Met
Number analyzed (Participants) | 134 | 132
mg/dL | -73.5 (4.055) | -38.0 (4.104)
Statistical Analysis 1: Comparison: Dapa+Saxa+Met vs Pla+Saxa+Met; Test type: Superiority or Other; p < 0.0001, Longitudinal Repeated Measures Analysis — Secondary end points are tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -35.5, 95% CI 2-sided [-46.3 to -24.7], Standard Error of Mean 5.493

4. Secondary Outcome: Adjusted Mean Change From Baseline in Body Weight at Week 24
Description: Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weights were measured during the qualification and lead-in periods and on Day 1 and Weeks 6, 12, 18, and 24 in the double-blind period.
Time Frame: From baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Dapa+Saxa+Met | Pla+Saxa+Met
Number analyzed (Participants) | 158 | 158
kg | -1.91 (0.2191) | -0.41 (0.2270)
Statistical Analysis 1: Comparison: Dapa+Saxa+Met vs Pla+Saxa+Met; Test type: Superiority or Other; p < 0.0001, Longitudinal Repeated Measures Analysis — Secondary endpoints are tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -1.50, 95% CI 2-sided [-2.12 to -0.89], Standard Error of Mean 0.3126

5. Secondary Outcome: Percentage of Subjects Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) <7.0% at Week 24 (Last Observation Carried Forward [LOCF])
Description: Percent adjusted for baseline HbA1c. Therapeutic glycemic response is defined as HbA1c <7.0%. Data after rescue medication was excluded from this analysis.
Time Frame: From baseline to week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Dapa+Saxa+Met | Pla+Saxa+Met
Number analyzed (Participants) | 158 | 158
Percentage of subjects | 36.7 | 13.3
Statistical Analysis 1: Comparison: Dapa+Saxa+Met vs Pla+Saxa+Met; Test type: Superiority or Other; p < 0.0001, Modified logistic regression — Secondary end points are tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = 25.5, 95% CI 2-sided [16.7 to 34.4]

ADVERSE EVENTS:
Groups:
- DAPA + SAXA + MET: Participants received dapagliflozin, 10 mg, and open-label saxagliptin 5 mg and metformin ≥1500 mg per day for up to 52 weeks
- PLA + SAXA + MET: Participants received dapagliflozin matching placebo and open-label saxagliptin 5 mg and metformin ≥1500 mg per day for up to 52 weeks
Arm/Group | DAPA + SAXA + MET | PLA + SAXA + MET
Serious Adverse Events (participants affected / at risk) | 7/160 | 4/160
Other Adverse Events (participants affected / at risk) | 103/160 | 112/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPA + SAXA + MET (N=160) | PLA + SAXA + MET (N=160)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
GANGRENE (Infections and infestations) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPA + SAXA + MET (N=160) | PLA + SAXA + MET (N=160)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (4) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 7 (7) | 9 (11)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 8 (9)
CHEST PAIN (General disorders) | 1 (1) | 4 (5)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 4 (4)
INFLUENZA (Infections and infestations) | 12 (14) | 12 (14)
NASOPHARYNGITIS (Infections and infestations) | 5 (5) | 8 (9)
PHARYNGITIS (Infections and infestations) | 6 (6) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 15 (19) | 16 (19)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 7 (9) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 5 (5) | 9 (10)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (10)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
DIZZINESS (Nervous system disorders) | 6 (6) | 0 (0)
HEADACHE (Nervous system disorders) | 11 (16) | 13 (15)
DEPRESSION (Psychiatric disorders) | 0 (0) | 5 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No